CLINICAL TRIAL: NCT01217658
Title: Measuring and Reducing Excessive Infant Crying: A Randomized Trial
Brief Title: Measuring and Reducing Excessive Infant Crying
Acronym: UTHealth THB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: National Institutes of Health (NIH) (NIH); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Christopher Greeley, Associate Professor - Pediatrics, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HSC-MS-10-0392; K23HD065872 (NIH)
Record Dates: First submitted 2010-10-06; First posted 2010-10-08 (Estimated); Last update posted 2015-12-08 (Estimated); Status verified 2015-12

CONDITIONS: Infant Colic; Postpartum Depression
Keywords: Randomized Trial; Infant Colic; Abusive Head Trauma; Shaken Baby Syndrome
MeSH Terms: conditions — Colic; Depression, Postpartum; Shaken Baby Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- The Happiest Baby on The Block (Experimental): Those receiving the intervention will be trained in the infant soothing techniques outlined in "The Happiest Baby on the Block".
  Interventions: Behavioral: The Happiest Baby on The Block
- AAP Education (Active Comparator): Those receiving the control group allocation will be counseled in the American Academy of Pediatrics guidelines regarding Infant Colic (AAP Infant Colic counseling).
  Interventions: Behavioral: AAP Infant Colic counseling

INTERVENTIONS:
Behavioral: The Happiest Baby on The Block — Those receiving the intervention will be trained in the infant soothing techniques outlined in "The Happiest Baby on the Block".
  Arms: The Happiest Baby on The Block
Behavioral: AAP Infant Colic counseling — Those receiving the control group allocation will be counseled using the American Academy of Pediatrics material for Infant Colic.
  Arms: AAP Education

SUMMARY:
Excessive infant crying (EIC) is likely to increase the risk of child abuse. The investigators propose a randomized trial using an intervention based on recommendations of Karp. The investigators will systematically identify 170 term infants with EIC and conduct assessments in the home at 6-8 weeks age to test the hypothesis that the intervention reduces mean infant hours of night-time crying, increases maternal soothing behaviors and improves parental anxiety and depression.

DETAILED DESCRIPTION:
Hypotheses: The soothing techniques taught to study parents 2-3 wks after birth augment parental soothing skills and reduces infant crying at night (primary outcome) and parental sleep loss, distress, & depression assessed in the home by a masked nurse at 8 wks.

Methods: Term singleton infants with EIC (> 3 hrs/24h) recruited through a program offered to parents at our hospital (4,700 births/yr) will be seen in our clinic 2-3 wks after birth. Consenting families (n=178) will be randomized to standard colic counseling (American Academy of Pediatrics) or to the intervention (adding nurse instruction plus a video and pamphlets). At 8 wks a study nurse will assess parental sleep and distress (Brief Symptom Inventory-18), place dosimeters in rooms where the infant sleeps and spends most time, and apply the actigraph at the ankle. She will collect the devices 5 days later, perform a physical exam at a usual feeding time (when EIC is likely), record infant & maternal behaviors during crying/feeding for the next 15 minutes using unobtrusive, validated methods (Tyson, 1992), and provide maternal support if desired. Standard statistical tests will be used (alpha=0.05; beta = 0.20; effect size =0.5 SD, power = .90).

ELIGIBILITY:
Inclusion Criteria:

* term, singleton neonates
* otherwise healthy
* parent must have at least a 6th grade understanding of English or Spanish
* infant must have colic (greater than 3 hours of crying per day)
* OR the infant's crying causes excessive stress on the either parent

Exclusion Criteria:

* cannot have a condition which would reasonably impact alertness or behavior

Ages: 3 Weeks to 5 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 28 (Actual)
Dates: Start 2011-01; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Mean night-time crying | 2 weeks after enrollment. Appproximately 6-8 weeks of life.
  Objectively recording night-time duration of excessive crying
Mean sleep duration | 2 weeks after enrollment. Appproximately 6-8 weeks of life.
  objectively measuring infant sleep duration

SECONDARY OUTCOMES:
Maternal Depression, Anxiety and Somatization | At study entry and conculsion (4 week interval); 2 weeks after enrollment. Appproximately 6-8 weeks of life.
  Using the BSI-18 at study enrollment and conclusion.
Salivary Biomarkers | At Study Entry and at 2 weeks after enrollment
  We are collecting maternal salivary cortisol and amylase at study entry and at study conclusion (within 2 weeks after enrollment)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Texas Health Science Center at Houston, Houston, Texas, United States

REFERENCES:
- See also: American Academy of Pediatrics Infant Colic Website — http://www.healthychildren.org/english/ages-stages/baby/crying-colic/Pages/default.aspx